CLINICAL TRIAL: NCT06252090
Title: Feasibility and Acceptability of Mentalization-based Treatment for Early Adolescents With Depression: A Short Term Psychotherapy Approach for Patients and Their Families
Brief Title: Feasibility and Acceptability Trial of a Short Term Mentalization Based Treatment for Adolescents With Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: University Diego Portales (Other)
Responsible Party: Principal Investigator, Javier Morán Kneer, Principal Investigator, Universidad de Valparaiso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEC 262-22
Record Dates: First submitted 2024-01-04; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Depression
Keywords: Depression; Adolescent; Mentalization; Family; Psychotherapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBT-A (Experimental): Short term Mentalization-based treatment for adolescents (psychotherapy).
  Interventions: Other: Short term mentalization-based treatment for adolescents (MBT-A)

INTERVENTIONS:
Other: Short term mentalization-based treatment for adolescents (MBT-A) — The general framework of intervention corresponds to the Mentalization-Based Treatment model for adolescents (MBT-A). In this study, the model was adapted to a brief, time-limited format (12 sessions) aimed at both the adolescent and their family. The model retains the main characteristics of Mentalization-Based Therapy, such as the therapist's basic attitude toward actively promoting patients' mentalization, uncertainty of mental states, focus on the here and now, and the use of affect as a mechanism for change.

SUMMARY:
A feasibility pilot trial that aims to evaluate the acceptability and feasibility of mentalization-based treatment for adolescents (MBT-A) adapted for early adolescents diagnosed with depression.

DETAILED DESCRIPTION:
Background. Adolescent depression is a highly prevalent public health concern, entailing substantial developmental impairments, a risk of chronicity, and severe outcomes, including suicide. Recent years have seen an escalation in depressive symptoms among adolescents, exacerbated by the COVID-19 pandemic. Currently, Chile lacks specific evidence-based clinical guidelines for family interventions in adolescent depression. Nonetheless, the executive summary of the Clinical Practice Guidelines for the Management of Adolescent Depression recognizes the need for such interventions. The 2022-2025 agenda for children and adolescents incorporates these interventions as part of the recommendations, addressing challenges identified by the System of Guarantees for the Comprehensive Protection of the Rights of Children and Adolescents and aligning with the International Convention on the Rights of Children and Adolescents' standards. The strategy proposed herein-a brief, mentalization-based treatment intervention for adolescents-aligns with two pivotal considerations for adolescent mental health care: accommodating the neurodevelopmental changes and vulnerabilities of this demographic, and leveraging the preventative potential of family interventions at a systemic level.

Aims. The study is a feasibility pilot trial that aims to evaluate the acceptability and feasibility of a short term mentalization based treatment for adolescents (MBT-A). 15 families of adolescents with a diagnosis of mild and moderate unipolar depression between 10 and 14 years old who consult at a primary health care center in Valparaíso will be recruited.

Methods. The design is based on the principles of the Consolidated Standards of Reporting Trials - Extension to Randomized Pilot and Feasibility Trials (CONSORT). Acceptability and feasibility outcomes will be assessed by means of questionnaires and interviews with both consultants and interveners, considering the training, clinical supervision, and intervention processes. Feasibility (recruitment, data attrition, and follow-up rates) and acceptability (adherence rate and CEQ) of the intervention, along with depressive (PHQ-9/RCADS-30), anxious (DASS-21), externalizing/internalizing (SDQ-SF) symptomatology, and Family Cohesion (FACES III) as secondary outcomes, will be considered. Therapeutic alliance (VTAS-SF), adherence to the therapeutic model (MBT-ACS), quality of patients' mentalization (OMP-A), and psychological well-being (CORE-OM/YP-CORE) will be assessed as well. The results of the analysis of interviews, as well as the calculation of the effect size of the intervention for the various outcomes, are considered as parameters and guidelines for a future RCT.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate major depressive disorder (DSM-5-TR and psychiatric interview).
* Written informed consent.
* Presence of at least one legally responsible adult consenting to participate in the therapeutic process.

Exclusion Criteria:

* Diagnoses of autism spectrum disorders
* Psychosis
* Bipolar affective disorder
* Active suicidal ideation
* Substance use disorder.
* Pregnancy

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | After 3 months (at the end of therapy)
  Number of subjects who agree to participate in the study compared to the number of subjects who are invited.
Data attrition rate | After 3 months (at the end of therapy)
  Number of subjects who complete the study with respect to subjects who are originally enrolled.
Follow-up rate | After 6 months (3 months after the end of therapy)
  Number of subjects completing treatment and completing follow-up evaluations
Adherence rate | After 3 months (at the end of therapy)
  Percentage of subjects completing all protocol assessments (including attendance at all 12 sessions).
Overall satisfaction with the intervention | Change from baseline in CEQ at 3 months (at the end of therapy)
  Credibility/Expectancy Questionnaire (CEQ). Values range between 0 and 10 points. Each of the 8 items are analyzed separately. Higher scores indicate a better outcome, with the exception of item 6, which is reversed.

SECONDARY OUTCOMES:
Depressive symptomatology (adolescents) | Change from baseline in the RCADS-30 depression subscale scores at 3 months (end of therapy) and at 5 months (follow-up)]
  Depression subscale of the Revised Child Anxiety and Depression Scale-30 (RCADS-30) for adolescents. Values range between 0 and 15 points. Lower scores indicate a better outcome.
Depressive symptomatology (responsible adult) | Change from baseline in PHQ-9 scores at 3 months (end of therapy) and 5 months (follow up).
  Patient Health Questionnaire-9 (PHQ-9). Values range between 0 and 27 points. Lower scores indicate a better outcome.
Anxious symptomatology (adolescent) | Change from baseline in Generalized anxiety subscale of the Revised Child Anxiety and Depression Scale-30 (RCADS-30) for adolescents scores at 3 months (end of therapy) and 5 months (follow up).
  Generalized anxiety subscale of the Revised Child Anxiety and Depression Scale-30 (RCADS-30) for adolescents. Values range between 0 and 15 points. Lower scores indicate a better outcome.
Anxious symptomatology (responsible adult) | Change from baseline in Anxiety subscale of the Depression, Anxiety and Stress Scale-21 (DASS-21) scores at 3 months (end of therapy) and 5 months (follow up).
  Anxiety subscale of the Depression, Anxiety and Stress Scale-21 (DASS-21). Values range between 0 and 21 points. Lower scores indicate a better outcome.
Externalizing and internalizing symptomatology (adolescent) | Change from baseline in the SDQ-SF scores at 3 months (end of therapy) and at 5 months (follow-up)
  Strengths and Difficulties Questionnaire - Short Form (SDQ-SF). Values range between 0 and 40 points. Lower scores indicate a better outcome.
Family cohesion | Change from baseline in the FACES III scores at 3 months (end of therapy) and at 5 months (follow-up)
  Family Cohesion (FACES III). Values range between 0 and 50 points. Values between 41 to 45 (cohesion) and 25 to 28 (adaptability) indicate a better outcome.

OTHER OUTCOMES:
Therapeutic alliance | Change in VTAS-SF scores through study completion, an average of 3 months
  Vanderbilt Therapeutic Alliance Scale - Short Form (VTAS-SF). Values range between 0 and 5 points. Each of the 5 items are analyzed separately. Higher scores indicate a better outcome, with the exception of item 3, which is reversed.
Adherence to the therapeutic model | Change in MBT-ACS scores through study completion, an average of 3 months
  Mentalization based treatment adherence and competence scale (MBT-ACS). Values range between 0 and 7 points. Higher scores indicate a better outcome.
Quality of patients' mentalization | Change in OMP-A scores through study completion, an average of 3 months
  Observational System for mentalization adolescent psychotherapy (OMP-A). Values range between 0 and 5 points. Higher scores indicate a better outcome.
Psychological well-being (responsible adult) | Change in CORE-OM through study completion, an average of 3 months
  Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM). Values range between 0 and 136 points. Lower scores indicate a better outcome.
Psychological well-being (adolescent) | Change in YP-CORE through study completion, an average of 3 months
  Young Person's Clinical Outcomes in Routine Evaluation (YP-CORE). Values range between 0 and 40 points. Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Jean & Marrie Thierry family public health center, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No